CLINICAL TRIAL: NCT06601543
Title: Predictors of Steroid Resistance in Pediatric Acute Immune Thrombocytopenic Purpura
Brief Title: Steroid Resistance in Pediatric Immune Thrombocytopenic Purpura
Acronym: ITP
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shereen Hassan abd Elrady Mohammed, Predictors of steroid resistance in pediatric acute immune thrombocytopenic purpura, Assiut University
Other Study IDs: Steroid resistance in ITP
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pediatric Mmune Thrombocytopenic Purpura

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To Predicting steroid resistance on children newly diagnosed with immune thrombocytopenic purpura

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP, platelet counts < 100 × 109/L) is the most common acquired childhood bleeding disorder, clinically characterized by a low platelet count in the absence of other thrombocytopenia causes [1,2].

The estimated incidence of ITP is 100 cases out of a million people per year; about half of these cases occur in previously healthy children, where it represents the most frequent blood disorder [3].

Most children present with a typical history of acute purpura and bruising after a mild viral infection [4]. In severe cases, intracranial hemorrhage (the most 0.5% serious complication, but also the rarest occurring in adults), gastrointestinal hemorrhage in 1.5 % of children, and genitourinary hemorrhage may occur [5].

The International Working Group on ITP defines ITP according to the following clinical phases [6]. These are as follows:

Newly diagnosed ITP is in the first three months post-diagnosis. Persistent ITP is for 3-12 months. Chronic ITP is for > 12 months. Refractory ITP is the failure to restore count of platelet after splenectomy. For children requiring therapy but without life threatening bleeding, corticosteroids are the recommended first line therapy over IVIG or anti-D [2].

Guidelines from the American Society of Hematology recommend a 5-7-day course of prednisone dosed at 2-4 mg/kg/day [2]. Seventy-five percent of children respond to steroids, with platelets recovering to hemostatic range by 2-7 days [7]. If a more rapid rise in platelets is desired, IV methylprednisolone may be used. Studies comparing outcomes between anti-D versus methylprednisolone [8] and comparing methylprednisolone with dexamethasone [9] showed similar response rates with minor side effects in all groups.

A study shows that 98% of patients with corticosteroid exposure experienced one or more side events, and 38% of patients need to stop or reduce corticosteroid therapy [10].

This research aims to develop a new prediction model to evaluate whether newly ITP patients are at high-risk of corticosteroid resistance, and help clinicians to choose better therapy so we divide patients to two groups, steroid response and steroid resistance.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed as acute immune thrombocytopenic purpura based on clinical manifestations and laboratory investigations from age of 1 years to age of 18 years.

Gender: both six

Exclusion Criteria:

* children with immune thrombocytopenic purpura below age of 1 years and above 18 years, patient with thrombocytopenic purpura with secondary causes, and chronic ITP

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children diagnosed ITP and take steroid an treatment
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
predicting steroid resistance on children with acute immune thrombocytopenic purpura in comparison between steroid resistant group and steroid sensitive group Secondary (subsidiary): | Baseline
  predicting steroid resistance on children with acute immune thrombocytopenic purpura in comparison between steroid resistant group and steroid sensitive group to allow early introduction of alternative therapy before bleeding symptoms occurs and to avoid side effects of steroid use.

CONTACTS AND LOCATIONS:
Overall Officials: Azza Ahmed El-Tayab, Principal Investigator; Mervat Amin Mahmoud, Study Director

REFERENCES:
- [Background] Buchanan GR, Adix L. Grading of hemorrhage in children with idiopathic thrombocytopenic purpura. J Pediatr. 2002 Nov;141(5):683-8. doi: 10.1067/mpd.2002.128547. PMID 12410198
- [Background] Su Y, Xu H, Xu Y, Yu J, Dai B, Xian Y, Xiao J. A retrospective analysis of therapeutic responses to two distinct corticosteroids in 259 children with acute primary idiopathic thrombocytopenic purpura. Hematology. 2009 Oct;14(5):286-9. doi: 10.1179/102453309X12473408860343. PMID 19843385
- [Background] Celik M, Bulbul A, Aydogan G, Tugcu D, Can E, Uslu S, Dursun M. Comparison of anti-D immunoglobulin, methylprednisolone, or intravenous immunoglobulin therapy in newly diagnosed pediatric immune thrombocytopenic purpura. J Thromb Thrombolysis. 2013 Feb;35(2):228-33. doi: 10.1007/s11239-012-0801-z. PMID 22956408
- [Background] Provan D, Stasi R, Newland AC, Blanchette VS, Bolton-Maggs P, Bussel JB, Chong BH, Cines DB, Gernsheimer TB, Godeau B, Grainger J, Greer I, Hunt BJ, Imbach PA, Lyons G, McMillan R, Rodeghiero F, Sanz MA, Tarantino M, Watson S, Young J, Kuter DJ. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood. 2010 Jan 14;115(2):168-86. doi: 10.1182/blood-2009-06-225565. Epub 2009 Oct 21. PMID 19846889
- [Background] Arnold DM. Bleeding complications in immune thrombocytopenia. Hematology Am Soc Hematol Educ Program. 2015;2015:237-42. doi: 10.1182/asheducation-2015.1.237. PMID 26637728
- [Background] Kuhne T, Buchanan GR, Zimmerman S, Michaels LA, Kohan R, Berchtold W, Imbach P; Intercontinental Childhood ITP Study Group; Intercontinental Childhood ITP Study Group. A prospective comparative study of 2540 infants and children with newly diagnosed idiopathic thrombocytopenic purpura (ITP) from the Intercontinental Childhood ITP Study Group. J Pediatr. 2003 Nov;143(5):605-8. doi: 10.1067/s0022-3476(03)00535-3. PMID 14615730
- [Background] Consolini R, Legitimo A, Caparello MC. The Centenary of Immune Thrombocytopenia - Part 1: Revising Nomenclature and Pathogenesis. Front Pediatr. 2016 Oct 19;4:102. doi: 10.3389/fped.2016.00102. eCollection 2016. PMID 27807534
- [Background] Neunert C, Terrell DR, Arnold DM, Buchanan G, Cines DB, Cooper N, Cuker A, Despotovic JM, George JN, Grace RF, Kuhne T, Kuter DJ, Lim W, McCrae KR, Pruitt B, Shimanek H, Vesely SK. American Society of Hematology 2019 guidelines for immune thrombocytopenia. Blood Adv. 2019 Dec 10;3(23):3829-3866. doi: 10.1182/bloodadvances.2019000966. PMID 31794604
- [Background] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182
- [Background] Zitek T, Weber L, Pinzon D, Warren N. Assessment and Management of Immune Thrombocytopenia (ITP) in the Emergency Department: Current Perspectives. Open Access Emerg Med. 2022 Jan 29;14:25-34. doi: 10.2147/OAEM.S331675. eCollection 2022. PMID 35125895
- See also: Related Info — https://www.hematology.org/